CLINICAL TRIAL: NCT02830802
Title: Randomized Controlled Clinical Trial for Evaluating a Sage-based Mouthrinse in Regard to Its Anti-inflammatory Potential in Elderly Patients Which Are Dependent in Their ADLs
Brief Title: Clinical Trial for Evaluating Sage-Based Mouthrinse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: WALA Heilmittel GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: gerodont_3: Sage Trial
Record Dates: First submitted 2016-07-01; First posted 2016-07-13 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Stomal Bleeding; Stomatitis, Denture; Tooth Staining; Satisfaction
MeSH Terms: conditions — Stomatitis, Denture; Tooth Discoloration; Personal Satisfaction | interventions — Cosmetics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Active Agent
  Interventions: Other: Dr. Hauschka Med Mundspüllösung Salbei / cosmetics
- Group B (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Dr. Hauschka Med Mundspüllösung Salbei / cosmetics — Supervised use over 6 weeks 1x/day additional to habitual oral hygiene protocol.
  For an application fill the closure cap with the mouthwash. Rinse the mouth vigorously for 30 seconds, for easier timekeeping use the hourglass. Then spit out the mouthwash, do not rinse.
  Arms: Group A
Other: Placebo — Supervised use over 6 weeks 1x/day additional to habitual oral hygiene protocol.
  For an application fill the closure cap with the mouthwash.
  Arms: Group B

SUMMARY:
The investigators aim to evaluate a sage-based mouthrinse (Dr. Hauschka Med, Mundspülung Salbei) whether it is less or equal effective in alleviating inflammatory signs of intra-oral mucosa and gingiva than an water/alcohol-based taste adjusted placebo in patients dependent on ADL.

Randomization in treatment A (mouthwash with active agent, n=24) or treatment B (placebo mouthwash, n=24) Supervised use of mouthwash A or mouthwash B over 6 weeks 1x/day additional to habitual oral hygiene protocol.

The main outcome parameter will be Sulcus Bleeding Index SBI.

DETAILED DESCRIPTION:
A sage-based mouthrinse based on an extract from Salvia officinalis in a composition with extracts from Althaea Officinalis, Aesculus Hippocatanum Bark and essential oils might comprise an alternative to conventional antimicrobial mouthrinses, which might exhibit important side effects. Thus the aim of the current study is to test the null-hypothesis H0:

A sage-based mouthrinse (Dr. Hauschka Med, Mundspülung Salbei, WALA Heilmittel GmbH, Dorfstraße 1, 73087 Bad Boll/Eckwälden, Germany) is less or equal effective in alleviating inflammatory signs of intra-oral mucosa and gingiva than an water/alcohol-based taste adjusted placebo.

The placebo and the sage-based mouthrinse will be manufactured according to EU-Kosmetik-Verordnung 1223/2009 and provided by WALA Heilmittel GmbH, Dorfstraße 1, 73087 Bad Boll/Eckwälden, Germany together with the necessary safety documentation. The placebo will be an alcohol/ water based solution with a similar taste to the tested mouthrinse.

The main outcome parameter will be Sulcus Bleeding Index SBI. Among others, the main secondary outcome parameters will be Oral Health Related Quality of Life as assessed with the OHIP-14 G questionnaire, the Xerostomia inventory and a Tooth staining index.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent, i.e. no legal guardian appointed
* Willing to participate
* Depended on their ADLs (IADL)(24)
* Sulcus Bleeding Index (SBI) > 50%

Exclusion Criteria:

* Allergy to one of the components
* Edentulous
* Alcohol dependency
* Prescription of antibiotics and/ or immunosuppressives (e.g. glucocorticoids) Anti-inflammatory mouthrinse -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-10; Primary Completion 2017-10 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Sulcus Bleeding Index | six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schimmel, Prof., Study Chair — University of Bern
Locations (1):
- University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No